CLINICAL TRIAL: NCT04052984
Title: Delayed Cord Clamping and Early Skin-to-skin Contact in Cesarean Section as Interventions That Promote Exclusive Breastfeeding
Brief Title: Interventions That Promote Exclusive Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asociacion Mexicana de Nacimiento Respetado, A.C. (Other)
Responsible Party: Principal Investigator, Farid Adán Pacheco Y Orozco, Investigator, Asociacion Mexicana de Nacimiento Respetado, A.C.
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 1
Record Dates: First submitted 2019-08-05; First posted 2019-08-12 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Breastfeeding, Exclusive
Keywords: Cesarean Section; Umbilical cord; Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: An intervention group compared to a similar historical group attended by the same group of doctors at an immediate previous time
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Twenty four pares of healthy mothers-newborns, with delayed clamping and immediate skin-to-skin contact after birth by caesarean section
  Interventions: Procedure: Delayed umbilical clamping and immediate skin-to-skin contact after birth by caesarean section
- Control group (No Intervention): Twenty four pares of healthy mothers-newborns, with early clamping without skin-to-skin contact after birth by caesarean section and newborn attended in radiant warm table

INTERVENTIONS:
Procedure: Delayed umbilical clamping and immediate skin-to-skin contact after birth by caesarean section — Mother: Placement of the insulating surgical arch was on the skin, between the abdomen and the thorax, electrocautery plate on the back, the gown superimposed, non-invasive blood pressure monitoring in legs and ear oximetry. The newborn was placed immediately on the mother's chest, passing it under the insulating arch and removing the mother's gown. Non-invasive monitoring was initiated with preductal pulse oximetry. The obstetrician cut the umbilical cord by not feeling the beats of the cord, or until 5 minutes. The newborn was reanimated without separating the baby from his mother. The temperature was taken with an infrared thermometer. Pulse oximetry was recorded. The newborn was colocated to the mother's breast as soon as possible, even if the mother was still in surgery. The mother's transfer to her room was with her baby skin to skin. The support staff was instructed not to separate the newborn until breast feeding occur for the first time or the mother required it.
  Arms: Intervention group

SUMMARY:
Delayed umbilical cord clamping as well as immediate skin-to-skin contact between mother and newborn are emerging practices due to documented benefits. However, in caesarean sections it is not common.

The investigators evaluate twenty four pares of healthy mothers-newborns, with delayed clamping and immediate skin-to-skin contact after birth by caesarean section (intervention grup), compared to the same number of pairs attended by the same group of physicians under traditional techniques (control group). In both groups, morbidity and mortality as well as sole breastfeeding was evaluated for at least 6 months. The patients in the intervention group signed an informed consent form and the protocol was approved by an ethics committee.

DETAILED DESCRIPTION:
BACKGROUND: Delayed umbilical cord clamping as well as immediate skin-to-skin contact between mother and newborn are emerging practices due to documented benefits for the mother-child binomial. The American Academy of Pediatrics, through the neonatal resuscitation program, considers that late clamping should be a common practice in all healthy babies, but in the case of a baby at risk, it recommends cutting the umbilical cord early and treating newborn on radiant warmer for resuscitation. Caesarean birth is considered a risk factor.

In Mexico and in many other countries early contact, skin to skin between the mother and child in Cesarean sections, is not common.

The World Health Organization (WHO), among multiple strategies to promote breastfeeding, promotes skin-to-skin contact at birth, that is: "to place babies with their mothers since birth minimal an hour or until the baby has been fed to the mother's breast". Different publications has determined that the ideal period to strengthen breastfeeding corresponds to the first minutes of life and does not go beyond the first 2 hours. Because it is usual to take care of the baby in radiant warmer, away from his mother, in caesarean sections, these recommendations are generally not met.

Searching the benefit of delayed cut of the umbilical cord, researchers began placing healthy babies in their mother's chest, even in cesarean deliveries, thus generating immediate skin-to-skin contact and incidentally an increase in the frequency of breastfeeding during the first six months, so a protocol was initiated to compare the morbidity and mortality of this technique in relation to traditional care (immediate cut of the umbilical cord and separation mother-child) and follow-up of babies at least six months to register the form of breastfeeding.

MATERIAL AND METHODS: Pilot study. All healthy mother-neonates binomials, obtained by caesarean section by the same medical team in 3 private hospitals, born between January 2015 and August 2017 in Villahermosa, Tabasco, Mexico followed for a minimum of 6 months in the private consultation were included. They were compared with an equal number of historical binomials, attended by the same medical team under the traditional technique and with the same follow-up time. The variables in this group were collected from their files.

By protocol of the medical group in both groups, it was encouraged to carry out an adequate program of exclusive breastfeeding, as marked by the World Health Organization consisting of starting breastfeeding in the first hour of life, that the Infant only received breast milk excluding other beverages such as water, teas or food, that breastfeeding was made on demand, as often as the child wanted both day and night and no bottles or pacifiers were used during his hospital stay.

The statistical evaluation included univariate analysis with frequencies and proportions for qualitative variables, measures of central tendency and dispersion for qualitative variables. In the bivariate analysis, X2 (or Fisher's Exact test) and Student's t (or Mann Whitney U) were used, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Controlled pregnancies
* Pregnancies not complicated
* Single product
* Signed the informed consent to participate in the protocol
* Product obtained by caesarean section.

Exclusion Criteria:

* Patients who did not wish to participate in the study
* Infants with prenatally suspected or diagnosticated congenital defects
* Multiple pregnancy
* Cases requesting to collect umbilical cord blood for storage in a cord cell bank
* Vaginal delivery

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Duration of feeding to the exclusive maternal breast | six months or more
  Time in months when the newborn was fed to the exclusive maternal breast

CONTACTS AND LOCATIONS:
Overall Officials: FARID ADAN PACHECO Y OROZCO, MD, Principal Investigator — Asociación Mexicana del Nacimiento Respetado

IPD SHARING:
Plan to Share IPD: Yes
All available data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: available data
Access Criteria: email

REFERENCES:
- [Background] Hutton EK, Hassan ES. Late vs early clamping of the umbilical cord in full-term neonates: systematic review and meta-analysis of controlled trials. JAMA. 2007 Mar 21;297(11):1241-52. doi: 10.1001/jama.297.11.1241. PMID 17374818
- [Background] Katheria AC, Brown MK, Faksh A, Hassen KO, Rich W, Lazarus D, Steen J, Daneshmand SS, Finer NN. Delayed Cord Clamping in Newborns Born at Term at Risk for Resuscitation: A Feasibility Randomized Clinical Trial. J Pediatr. 2017 Aug;187:313-317.e1. doi: 10.1016/j.jpeds.2017.04.033. Epub 2017 May 16. PMID 28526223
- [Background] Vatansever B, Demirel G, Ciler Eren E, Erel O, Neselioglu S, Karavar HN, Gundogdu S, Ulfer G, Bahadir S, Tastekin A. Is early cord clamping, delayed cord clamping or cord milking best? J Matern Fetal Neonatal Med. 2018 Apr;31(7):877-880. doi: 10.1080/14767058.2017.1300647. Epub 2017 Mar 20. PMID 28320218
- [Background] Koopman I, Callaghan-Koru JA, Alaofin O, Argani CH, Farzin A. Early skin-to-skin contact for healthy full-term infants after vaginal and caesarean delivery: a qualitative study on clinician perspectives. J Clin Nurs. 2016 May;25(9-10):1367-76. doi: 10.1111/jocn.13227. Epub 2016 Mar 30. PMID 27027262
- [Background] Stevens J, Schmied V, Burns E, Dahlen H. Immediate or early skin-to-skin contact after a Caesarean section: a review of the literature. Matern Child Nutr. 2014 Oct;10(4):456-73. doi: 10.1111/mcn.12128. Epub 2014 Apr 10. PMID 24720501
- [Background] Wyckoff MH, Aziz K, Escobedo MB, Kapadia VS, Kattwinkel J, Perlman JM, Simon WM, Weiner GM, Zaichkin JG. Part 13: Neonatal Resuscitation: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care (Reprint). Pediatrics. 2015 Nov;136 Suppl 2:S196-218. doi: 10.1542/peds.2015-3373G. Epub 2015 Oct 14. No abstract available. PMID 26471383
- [Background] Kumar P, Yamada NK, Fuerch JH, Halamek LP. The neonatal resuscitation program: current recommendations and a look at the future. Indian J Pediatr. 2014 May;81(5):473-80. doi: 10.1007/s12098-013-1332-0. Epub 2014 Mar 22. PMID 24652267
- [Background] Kollmann M, Aldrian L, Scheuchenegger A, Mautner E, Herzog SA, Urlesberger B, Raggam RB, Lang U, Obermayer-Pietsch B, Klaritsch P. Early skin-to-skin contact after cesarean section: A randomized clinical pilot study. PLoS One. 2017 Feb 23;12(2):e0168783. doi: 10.1371/journal.pone.0168783. eCollection 2017. PMID 28231274
- [Background] Brimdyr K, Cadwell K, Stevens J, Takahashi Y. An implementation algorithm to improve skin-to-skin practice in the first hour after birth. Matern Child Nutr. 2018 Apr;14(2):e12571. doi: 10.1111/mcn.12571. Epub 2017 Dec 12. PMID 29230957
- [Background] Moore ER, Bergman N, Anderson GC, Medley N. Early skin-to-skin contact for mothers and their healthy newborn infants. Cochrane Database Syst Rev. 2016 Nov 25;11(11):CD003519. doi: 10.1002/14651858.CD003519.pub4. PMID 27885658
- [Background] World Health Organization Human Reproduction Programme, 10 April 2015. WHO Statement on caesarean section rates. Reprod Health Matters. 2015 May;23(45):149-50. doi: 10.1016/j.rhm.2015.07.007. Epub 2015 Jul 27. No abstract available. PMID 26278843
- [Background] Gomez Papi A, Baiges Nogues MT, Batiste Fernandez MT, Marca Gutierrez MM, Nieto Jurado A, Closa Monasterolo R. [Kangaroo method in delivery room for full-term babies]. An Esp Pediatr. 1998 Jun;48(6):631-3. Spanish. PMID 9662849
- [Background] Beake S, Bick D, Narracott C, Chang YS. Interventions for women who have a caesarean birth to increase uptake and duration of breastfeeding: A systematic review. Matern Child Nutr. 2017 Oct;13(4):e12390. doi: 10.1111/mcn.12390. Epub 2016 Nov 24. PMID 27882659
- [Background] Diaz-Castro J, Florido J, Kajarabille N, Garrido-Sanchez M, Padilla C, de Paco C, Navarrete L, Ochoa JJ. The timing of cord clamping and oxidative stress in term newborns. Pediatrics. 2014 Aug;134(2):257-64. doi: 10.1542/peds.2013-3798. Epub 2014 Jul 14. PMID 25022744
- [Background] Hooper SB, Binder-Heschl C, Polglase GR, Gill AW, Kluckow M, Wallace EM, Blank D, Te Pas AB. The timing of umbilical cord clamping at birth: physiological considerations. Matern Health Neonatol Perinatol. 2016 Jun 13;2:4. doi: 10.1186/s40748-016-0032-y. eCollection 2016. PMID 27298730
- [Background] van Rheenen PF, Brabin BJ. A practical approach to timing cord clamping in resource poor settings. BMJ. 2006 Nov 4;333(7575):954-8. doi: 10.1136/bmj.39002.389236.BE. No abstract available. PMID 17082547